CLINICAL TRIAL: NCT02519699
Title: Microcirculation After MAP Increase in Septic Shock Patients With Previous Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Flavia Ribeiro Machado, Professor and Chair of Intensive Care Anesthesiology, Pain and Intensive Care Department, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEP173.166
Record Dates: First submitted 2015-07-28; First posted 2015-08-11 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Norepinephrine (Experimental): Noradrenaline continuous infusion IV
  Interventions: Drug: norepinephrine

INTERVENTIONS:
Drug: norepinephrine — Increase in mean arterial pressure using norepinephrine
  Other Names: noradrenaline

SUMMARY:
The optimal levels of mean arterial pressure that must be achieved in septic shock are subject of debate. Studies tried to correlate blood pressure increase in patients with septic shock with microcirculation. However, there are few studies that specifically assessed septic shock patients with previous arterial hypertension. The main objective of this study is to evaluate the effect of increased blood pressure level in the microcirculation of these patients and compare them with patients without arterial hypertension.

DETAILED DESCRIPTION:
Hypothesis: After a rise in mean arterial pressure, microcirculation improvement will occur only in the previously hypertensive patients.

Study design: Prospective clinical trial Setting: Intensive care units of the Anesthesiology Department at the Federal University of Sao Paulo and the intensive care unit of Kidney Hospital.

Studied population: Forty patients will be included, being 20 without known history of systemic arterial hypertension and 20 with this diagnosis for at least 2 years and already with clinical or subclinical organ damage.

Inclusion criteria: age over than 18 years old, norepinephrine drug use for at least 12 hours and for less than 72 hours, sedation level equal or deeper than Ramsay 4, blood pressure stable for the last 30 minutes prior to inclusion, central venous catheter in place and signed informed consent.

Exclusion criteria: pregnancy, cirrhosis, systemic sclerosis, and need to maintain mean arterial pressure above 65mmHg for others conditions.

Intervention: noradrenaline dose will be risen to obtain a mean arterial pressure of 85-90 mmHg.

Assessments and outcome: Systemic hemodynamic (central venous oxygen saturation, cardiac output, heart rate, central venous pressure) and sublingual microcirculation variables (microcirculatory flow index, total vascular density, proportion of perfused vessels, perfused vascular density) will be measured before and after the rise in mean arterial pressure. Sidestream darkfield will be used to assess microcirculation. The variation between those variables before and after the intervention will be compared.

ELIGIBILITY:
Inclusion Criteria:

* age over than 18 years old,
* norepinephrine drug use for at least 12 hours and for less than 72 hours,
* sedation level equal or deeper than Ramsay 4,
* blood pressure stable for the last 30 minutes prior to inclusion,
* central venous catheter in place and
* signed informed consent.

Exclusion Criteria:

* pregnancy,
* cirrhosis,
* systemic sclerosis, and
* need to maintain mean arterial pressure above 65mmHg for others conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Microcirculatory flow index (MIF) measured by sidestream darkfield after rising the mean arterial pressure with norepinephrine | after 20 min
  MIF will be measured in points varying from 0 to 4

SECONDARY OUTCOMES:
Total vascular density (TVD) measured by sidestream darkfield after rising the mean arterial pressure with norepinephrine | after 20 min
  TVD will be measured in mm/mm2
Perfused vascular density (PVD) measured by sidestream darkfield after rising the mean arterial pressure with norepinephrine | after 20 min
  PVD will be measured in mm/mm2
Proportional perfused vessels (PPV) measured by sidestream darkfield after rising the mean arterial pressure with norepinephrine | after 20 min
  PPV will be measured in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Machado, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Hospital São Paulo - Universidade Federal de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Background] Xu JY, Ma SQ, Pan C, He HL, Cai SX, Hu SL, Liu AR, Liu L, Huang YZ, Guo FM, Yang Y, Qiu HB. A high mean arterial pressure target is associated with improved microcirculation in septic shock patients with previous hypertension: a prospective open label study. Crit Care. 2015 Mar 30;19(1):130. doi: 10.1186/s13054-015-0866-0. PMID 25887027
- [Background] Dubin A, Pozo MO, Casabella CA, Palizas F Jr, Murias G, Moseinco MC, Kanoore Edul VS, Palizas F, Estenssoro E, Ince C. Increasing arterial blood pressure with norepinephrine does not improve microcirculatory blood flow: a prospective study. Crit Care. 2009;13(3):R92. doi: 10.1186/cc7922. Epub 2009 Jun 17. PMID 19534818
- [Background] Correa TD, Vuda M, Takala J, Djafarzadeh S, Silva E, Jakob SM. Increasing mean arterial blood pressure in sepsis: effects on fluid balance, vasopressor load and renal function. Crit Care. 2013 Jan 30;17(1):R21. doi: 10.1186/cc12495. PMID 23363690
- [Background] Leone M, Asfar P, Radermacher P, Vincent JL, Martin C. Optimizing mean arterial pressure in septic shock: a critical reappraisal of the literature. Crit Care. 2015 Mar 10;19(1):101. doi: 10.1186/s13054-015-0794-z. PMID 25888071
- [Derived] Fiorese Coimbra KT, de Freitas FGR, Bafi AT, Pinheiro TT, Nunes NF, de Azevedo LCP, Machado FR. Effect of Increasing Blood Pressure With Noradrenaline on the Microcirculation of Patients With Septic Shock and Previous Arterial Hypertension. Crit Care Med. 2019 Aug;47(8):1033-1040. doi: 10.1097/CCM.0000000000003795. PMID 31094744